CLINICAL TRIAL: NCT01517464
Title: A Phase I Study of Systemic Gene Therapy With SGT-94 in Patients With Solid Tumors
Acronym: SGT94-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SynerGene Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGT94-01
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Neoplasm
Keywords: neoplasm; bladder cancer; advances solid tumors
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SGT-94 (Experimental): Dose escalation of experimental therapeutic SGT-94 to assess safety
  Interventions: Genetic: SGT-94

INTERVENTIONS:
Genetic: SGT-94 — SGT-94 will be given at doses of 0.6, 1.2, 2.4, 3.6 and 4.8 mgDNA/infusion(Doses 0-5, respectively)twice weekly for 3 weeks out of 4 in dose levels 0 to 4, and for 5 weeks out of 6 for dose level 5 (also 4.8mg DNA). Intravenous infusion will occur over 1 to 2.5 hours in 5% dextrose,with a final volume of SGT-94 and dextrose of 100 mL to 250 mL, depending on dose level.

SUMMARY:
This is a Phase I study designed to evaluate the safety and maximum tolerated dose (MTD) of SGT-94, a novel, tumor-targeted, systemic gene therapy agent for cancer. In addition, we will look for evidence of RB94 expression within tumor tissue after systemic administration of SGT-94.

DETAILED DESCRIPTION:
RB94, a tumor suppressor gene, is a modified form of the retinoblastoma gene, RB110. RB94 has shown enhanced tumor suppressor and tumor cell killing activity compared to RB110 in all tumor cell types studied to date, including bladder cancer cell lines. Moreover, RB94 has shown no toxicity to any normal human cells tested.

SGT-94,the agent being tested, is a systemically administered complex composed of the RB94 gene (plasmid DNA)encapsulated in a liposome that is targeted to tumor cells by means of an anti-transferrin receptor single chain antibody fragment (TfRscFv)attached to the outside of the liposome. Pre-clinical in vivo efficacy studies have indicated that SGT-94, when systemically administered, preferentially targets tumor cells and efficiently transfects them. This results in cancer cell death via mechanisms that are unique for RB94 and also increases the tumor's response to conventional radiation and chemotherapy.

This Phase I study is designed to evaluate the safety of SGT-94 and to establish a practically attainable and/or tolerable dose of this anti-cancer agent for use in further clinical trials. Additionally, evidence of RB94 expression within tumor tissue after systemic administration of SGT-94 will be sought, and clinically observable anti-cancer effects in patients will be documented. Enrollment will be targeted to individuals with "RB negative" tumors, i.e. tumors in which there is no staining for RB protein by immunohistochemistry (IHC). Preference will be given to patients with tumors in a location amenable to biopsy following treatment with SGT-94. This would include the prostate, bladder, superficial lymph nodes and any mass suitable for fine needle aspiration under CT or ultrasound guidance, or any lesion reachable by endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer for which no standard therapy is available, and which shows no staining for RB by IHC.
* Spirometry with at least 70% of predicted volumes (including FEV1). A left ventricular ejection fraction (LVEF) of 45% or more. All patients will have a screening 2-D Echocardiogram as part of eligibility screening.
* Patients must have adequate physiologic reserve as evidenced by:

  * Zubrod Performance Status (PS) of </= 2; or 3 if of recent onset (i.e. < 2 weeks) and if the compromised performance status is related to uncontrolled pain which is expected to come under control by means of improved pain management.
  * Laboratory values meeting the following criteria:

    * Absolute neutrophil count >/= 1,200/mm3
    * Platelet count >100,000/mm3.
    * AST and ALT </= 3x the upper limit of normal
    * Conjugated bilirubin </= 1.5 mg/dL (or total bilirubin </= 2.5 mg/dL)
    * Native kidney function producing creatinine clearance (either measured or estimated by Cockcroft formula) of at least 40 mL/min. Cockcroft formula: CLcr = [(140-age) • wt(kg)]/[72 •Creat (mg/dL)] (For females, multiply by 0.85)
    * Hemoglobin >/= 10.0 g/dL without transfusion support
    * White blood cell count > 3.0 k/mm3
    * PT and aPTT each < 1.5 times the upper limit of normal.
* Women of child-bearing potential must have a negative pregnancy test.
* Male and female patients reproductive potential must agree to use measures to avoid pregnancy throughout the study and for 3 months following discontinuing study drug.
* Patients must have recovered from any previous therapy side effects or toxicities prior to initiating protocol study infusions.
* Life expectancy > 12 weeks.
* Organ function </= grade 1.
* Age of </= 18 years.

Exclusion Criteria:

* Some prior cancer therapies are not consistent with eligibility; specifically:

  * At least 30 days must have elapsed since any prior experimental therapy
  * At least 6 weeks must have elapsed since prior systemic mitomycin C
  * At least 8 weeks must have elapsed since any dose of Strontium-89
  * At least 4 weeks must have elapsed since prior Sm-153 lexidronam (Quadramet™)
  * At least 4 weeks must have elapsed since prior radiotherapy
  * Any prior exposure to gene vector delivery products
* Pregnancy or lactation
* Serious concurrent medical illness that in the opinion of the investigator would compromise patient safety or preclude accurate assessment of outcome.
* Patients with the following manifestations of cardiovascular disease are excluded:

  * Myocardial infarction (MI) within the previous six months, or patients with left ventricular ejection fraction of less than 45% secondary to a more remote MI.
  * Any history of CVA or TIA in previous six months
  * New York Heart Association grade 2 or greater congestive failure
  * Unstable angina defined as angina (or anginal equivalent) 2 or more times per week despite medical therapy.
  * Echocardiographic evidence of pulmonary hypertension.
  * Diastolic dysfunction felt to contribute to any clinical sign or symptom.
  * Uncontrolled hypertension, defined as systolic BP >140 or diastolic >90 despite therapy.
* Serious concurrent psychiatric disorder that in the opinion of the investigator would compromise patient safety or preclude accurate assessment of outcome.
* Supraphysiologic doses of glucocorticoids (defined as > 30 mg of hydrocortisone per day or > 7.5 mg of Prednisone per day, or equivalent doses of other agents) or exposure to other immunosuppressive medications in the previous 30 days.
* Requirement for anticoagulant therapy other than low intensity treatment to maintain patency of central venous catheters.
* Treatment with antibiotics for proven infection within 1 week prior to study entry or signs and symptoms consistent with an active infection or fever > 38.1 C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Severity of Adverse Events | 4 weeks each patient
  The severity of adverse experiences in each patient will be determined based upon changes in the results of clinical laboratory tests and physical examnations. These findings will be used to determine the safety and tolerability of increasing doses of SGT-94.

SECONDARY OUTCOMES:
Clinical Response | Week 4
  Clinical Response will be assessed according to standard criteria for the particular solid tumor. In general, Response Evaluation Criteria in Solid Tumors (RECIST) criteria will be used.
Changes in Tumor Markers | Week 4
  When appropriate, changes in tumor markers between the values measured at baseline and at week 4 following the cycle of SGT-94 infusion will be assessed.
Expression of RB94 in Tumor Biopsies | Week 2
  Tumor targeting and uptake of SGT-94 by the tumor cells will be determined using Immunohistochemistry to assess the expression of RB94 in any tumor biopsies obtained during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Siefker-Radtke, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas, M.D. Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pirollo KF, Rait A, Zhou Q, Zhang XQ, Zhou J, Kim CS, Benedict WF, Chang EH. Tumor-targeting nanocomplex delivery of novel tumor suppressor RB94 chemosensitizes bladder carcinoma cells in vitro and in vivo. Clin Cancer Res. 2008 Apr 1;14(7):2190-8. doi: 10.1158/1078-0432.CCR-07-1951. PMID 18381961
- [Background] Xu HJ, Xu K, Zhou Y, Li J, Benedict WF, Hu SX. Enhanced tumor cell growth suppression by an N-terminal truncated retinoblastoma protein. Proc Natl Acad Sci U S A. 1994 Oct 11;91(21):9837-41. doi: 10.1073/pnas.91.21.9837. PMID 7937901
- [Background] Xu HJ, Zhou Y, Seigne J, Perng GS, Mixon M, Zhang C, Li J, Benedict WF, Hu SX. Enhanced tumor suppressor gene therapy via replication-deficient adenovirus vectors expressing an N-terminal truncated retinoblastoma protein. Cancer Res. 1996 May 15;56(10):2245-9. PMID 8625292
- [Background] Zhou J, Zhang XQ, Ashoori F, McConkey DJ, Knowles MA, Dong L, Benedict WF. Early RB94-produced cytotoxicity in cancer cells is independent of caspase activation or 50 kb DNA fragmentation. Cancer Gene Ther. 2009 Jan;16(1):13-9. doi: 10.1038/cgt.2008.54. Epub 2008 Jul 25. PMID 18654611